CLINICAL TRIAL: NCT03430063
Title: A Randomized, Open-Label Study of Combinations of Standard and High Dose REGN2810 (Cemiplimab; Anti-PD-1 Antibody) and Ipilimumab (Anti-CTLA-4 Antibody) in the Second-Line Treatment of Patients With Advanced Non-Small Cell Lung Cancer
Brief Title: A Study of REGN2810 and Ipilimumab in Patients With Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Business decision
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R2810-ONC-1763; 2017-003684-35 (EudraCT Number)
Record Dates: First submitted 2018-01-29; First posted 2018-02-12 (Actual); Results first posted 2022-11-03 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-10

CONDITIONS: Advanced Non-Small Cell Lung Carcinoma
Keywords: Advanced non-squamous NSCLC; Advanced squamous NSCLC
MeSH Terms: interventions — cemiplimab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- SDREGN2810 (Experimental)
  Interventions: Drug: SDREGN2810
- SDREGN2810/ipi (Experimental)
  Interventions: Drug: SDREGN2810/ipi
- HDREGN2810 (Experimental)
  Interventions: Drug: HDREGN2810

INTERVENTIONS:
Drug: SDREGN2810 — Standard dose intravenous (IV) infusion
  Other Names: REGN2810; cemiplimab
  Arms: SDREGN2810
Drug: SDREGN2810/ipi — Combination therapy dose IV
  Other Names: REGN2810; cemiplimab; ipilimumab
  Arms: SDREGN2810/ipi
Drug: HDREGN2810 — High dose IV
  Other Names: REGN2810; cemiplimab
  Arms: HDREGN2810

SUMMARY:
The primary objective of the study is to compare the objective response rate (ORR) of high dose cemiplimab (HDREGN2810) and standard dose cemiplimab plus ipilimumab combination therapy (SDREGN2810/ipi) to the ORR of standard dose cemiplimab (SDREGN2810) in the second-line treatment of patients with advanced squamous or non-squamous non-small cell lung cancer (NSCLC), in patients whose tumors express programmed cell death ligand 1 (PD-L1) in <50% of tumor cells.

ELIGIBILITY:
Key Inclusion Criteria:

1. Patients with histologically or cytologically documented squamous or non-squamous NSCLC who either have stage IIIb or stage IIIc disease who are not candidates for treatment with definitive concurrent chemo-radiation or have stage IV disease. Patients must have PD after receiving one prior line of chemotherapy treatment for advanced NSCLC.
2. Availability of an archival or on-study obtained formalin-fixed, paraffin-embedded tumor tissue biopsy sample
3. Biopsy evaluable for expression of PD-L1 as determined by a PD-L1 Immunohistochemistry (IHC) pharma diagnostic test (pharmDx) assay performed by a central laboratory
4. At least 1 radiographically measureable lesion by computed tomography (CT) per RECIST 1.1 criteria
5. Eastern Cooperative Oncology Group (ECOG) performance status of ≤1

Key Exclusion Criteria:

1. Patients who have never smoked, defined as smoking ≤100 cigarettes in a lifetime
2. Active or untreated brain metastases or spinal cord compression
3. Patients with tumors tested positive for epidermal growth factor receptor (EGFR) gene mutations, anaplastic lymphoma kinase (ALK) gene translocations, or C-ros oncogene receptor tyrosine kinase (ROS1) fusions
4. Encephalitis, meningitis, or uncontrolled seizures in the year prior to randomization
5. History of interstitial lung disease (eg, idiopathic pulmonary fibrosis or organizing pneumonia), or active, noninfectious pneumonitis that required immune-suppressive doses of glucocorticoids to assist with management, or of pneumonitis within the last 5 years
6. Ongoing or recent evidence of significant autoimmune disease that required treatment with systemic immunosuppressive treatments, which may suggest a risk of immunerelated treatment-emergent adverse events (irTEAEs)
7. Patients with a condition requiring corticosteroid therapy (>10 mg prednisone/day or equivalent) within 14 days of randomization

Note: Other protocol defined Inclusion/Exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2018-05-29 (Actual); Primary Completion 2021-10-27 (Actual); Study Completion 2021-10-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (29):
- United States (6):
  - Regeneron Research Site, Phoenix, Arizona
  - Regeneron Research Site, Los Angeles, California
  - Regeneron Research Site, Whittier, California
  - Regeneron Research Site, Scarborough, Maine
  - Regeneron Research Site, Canton, Ohio
  - Regeneron Research Site, Massillon, Ohio
- Belgium (2):
  - Regeneron Research Site, Herstal
  - Regeneron Research Site, Yvoir
- France (3):
  - Regeneron Research Site, Poitiers
  - Regeneron Research Site, Rennes
  - Regeneron Research Site, Saint-Mandé
- Regeneron Research Site, Gauting, Germany
- Poland (3):
  - Regeneron Research Site, Gdynia
  - Regeneron Research Site, Grudziądz
  - Regeneron Research Site, Otwock
- South Korea (5):
  - Regeneron Research Site, Incheon
  - Regeneron Research Site, Jeongnam
  - Regeneron Research Site, Seongnam
  - Regeneron Research Site, Seoul
  - Regeneron Research Site, Suwon
- Spain (5):
  - Regeneron Research Site, Badalona
  - Regeneron Research Site, Barcelona
  - Regeneron Research Site, Madrid
  - Regeneron Research Site, Málaga
  - Regeneron Research Site, Zaragoza
- Regeneron Research Site, Taipei, Taiwan
- United Kingdom (3):
  - Regeneron Research Site, London
  - Regeneron Research Site, Manchester
  - Regeneron Research Site, Plymouth

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Due to early enrollment cessation, only 28 participants were randomized and 27 participants received study treatment in this study. One participant was randomized but not treated.
Pre-assignment Details: Of the 27 participants treated, four participants completed the study. The most common reason for study discontinuation was death (8 participants) followed by withdrawal of consent (6 participants), and progressive disease (4 participants).
Groups:
- Cemiplimab 350 mg Q3W: Participants received 350 mg of cemiplimab intravenous (IV) infusion on Day 1 of every 3 weeks (Q3W) for up to 108 weeks or until progression of disease or unacceptable toxicity, withdrawal of consent, death, initiation of another anti-cancer treatment.
- Cemiplimab 350 mg Q3W + Ipilimumab 50 mg Q6W: Participants received 350 mg of cemiplimab IV infusion on Day 1 of Q3W for up to 108 weeks followed by ipilimumab 50 mg flat dose administered IV on Day 1 of every other treatment cycle (every 42 days or every 6 weeks [Q6W]) for up to 4 doses or until progression of disease or unacceptable toxicity, withdrawal of consent, death, initiation of another anti-cancer treatment.
- Cemiplimab 1050 mg Q3W: Participants received 1050 mg of cemiplimab IV infusion on Day 1 of Q3W for up to 108 weeks or until progression of disease or unacceptable toxicity, withdrawal of consent, death, initiation of another anti-cancer treatment.
Period: Overall Study
Arm/Group | Cemiplimab 350 mg Q3W | Cemiplimab 350 mg Q3W + Ipilimumab 50 mg Q6W | Cemiplimab 1050 mg Q3W
Started (All randomized participants) | 8 | 11 | 9
Treated (All randomized participants who received any study treatment) | 8 | 11 | 8
Completed (Completed study) | 0 | 3 | 1
Not Completed | 8 | 8 | 8
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Death | 3 | 2 | 3
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Withdrawal of consent | 3 | 1 | 2
Not completed — Progressive disease | 1 | 2 | 1
Not completed — Other un-specified | 1 | 1 | 0
Not completed — Randomized, but never treated | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety analysis set (SAF) included all randomized participants who received any study drug; it is based on the treatment received (as treated).
Groups:
- Cemiplimab 350 mg Q3W: Participants received 350 mg of cemiplimab IV infusion on Day 1 of Q3W for up to 108 weeks or until progression of disease or unacceptable toxicity, withdrawal of consent, death, initiation of another anti-cancer treatment.
- Total: Total of all reporting groups
Arm/Group | Cemiplimab 350 mg Q3W | Cemiplimab 350 mg Q3W + Ipilimumab 50 mg Q6W | Cemiplimab 1050 mg Q3W | Total
Number analyzed (Participants) | 8 | 11 | 8 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.4 (7.91) | 68.5 (8.72) | 68.1 (12.08) | 66.6 (9.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 1 | 7
  Male | 6 | 7 | 7 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 7 | 6 | 19
  Unknown or Not Reported | 2 | 4 | 2 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 6 | 3 | 3 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 5 | 3 | 8
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 3 | 2 | 7
Number of Participants with PD-L1 Tumor Expression Levels of ≥50% of Tumor Cells [Count of Participants; unit: Participants] — Number of participants with programmed death-ligand 1 (PD-L1) tumor expression levels of ≥50% of tumor cells is reported
  Participants | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) in Participants Whose Tumors Express Programmed Cell Death Ligand 1 (PD-L1) in <50% of Tumor Cells
Description: ORR was defined as the number of participants with a best overall response (BOR) of complete response (CR) or partial response (PR) divided by the number of participants in the efficacy analysis set. BOR was defined as the best response recorded, as determined by a blinded Independent Review Committee (IRC) based on Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) between the date of randomization and the date of the first objectively documented progression or the date of subsequent anti-cancer therapy, whichever came first. CR was defined as the disappearance of all target lesions (Any pathological lymph nodes [whether target or non-target] must have reduction in short axis to <10 mm [<1 cm]). PR was defined as having at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From date of randomization up to 41 months
Population: SAF included all randomized participants who received any study drug; it is based on the treatment received (as treated).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cemiplimab 350 mg Q3W | Cemiplimab 350 mg Q3W + Ipilimumab 50 mg Q6W | Cemiplimab 1050 mg Q3W
Number analyzed (Participants) | 8 | 11 | 8
Percentage of participants | 0 [0.0 to 36.9] | 45.5 [16.7 to 76.6] | 0 [0.0 to 36.9]

2. Secondary Outcome: Overall Response Rate
Description: Overall Response Rate was defined as the number of participants with a best overall response (BOR) of complete response (CR) or partial response (PR) divided by the number of participants in the efficacy analysis set. BOR was defined as the best response recorded, as determined by a blinded Independent Review Committee (IRC) based on Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) between the date of randomization and the date of the first objectively documented progression or the date of subsequent anti-cancer therapy, whichever came first. CR was defined as the disappearance of all target lesions (Any pathological lymph nodes [whether target or non-target] must have reduction in short axis to <10 mm [<1 cm]). PR was defined as having at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From date of randomization up to 41 months
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Cemiplimab 350 mg Q3W | Cemiplimab 350 mg Q3W + Ipilimumab 50 mg Q6W | Cemiplimab 1050 mg Q3W
Number analyzed (Participants) | 8 | 11 | 8
Percentage of participants
  Complete Response | 0 | 0 | 0
  Partial Response | 0 | 45.5 | 0

3. Secondary Outcome: Overall Survival (OS) in Participants With Tumor PD-L1 Expression Levels <50% of Tumor Cells
Description: OS was defined as the time from randomization to the date of death due to any cause. A participant who lost to follow-up was censored at the last date that the participant was known to be alive. OS was measured using Kaplan-Meier method.
Time Frame: Time from randomization to the date of death (up to 41 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cemiplimab 350 mg Q3W | Cemiplimab 350 mg Q3W + Ipilimumab 50 mg Q6W | Cemiplimab 1050 mg Q3W
Number analyzed (Participants) | 8 | 11 | 8
Months | 5.1 [1.7 to NA] — Data could not be estimated due to higher number (>50%) of censored participants. | NA [2.2 to NA] — Data could not be estimated due to higher number (>50%) of censored participants. | 8.4 [1.4 to NA] — Data could not be estimated due to higher number (>50%) of censored participants.

4. Secondary Outcome: Progression Free Survival (PFS) in Participants With Tumor PD-L1 Expression Levels <50% of Tumor Cells
Description: PFS was defined as the time from randomization to the date of the first documented tumor progression, as determined by the IRC (based on RECIST 1.1 assessments) or death due to any cause, whichever occurred earlier. PFS was measured using Kaplan-Meier method.
Time Frame: Time from randomization up to the date of the first documented tumor progression or death (up to 41 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cemiplimab 350 mg Q3W | Cemiplimab 350 mg Q3W + Ipilimumab 50 mg Q6W | Cemiplimab 1050 mg Q3W
Number analyzed (Participants) | 8 | 11 | 8
Months | 2.0 [0.7 to 8.3] | 20.8 [1.2 to NA] — Upper limit of 95% CI was not estimable due to low number of events. | 1.8 [1.1 to 2.2]

5. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs), Serious TEAEs, and TEAEs Resulting in Death
Description: Adverse event (AE): any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of study drug, whether or not considered related to the study drug. Serious AE: an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. TEAE: AE with onset after start of treatment or with onset date before the treatment start date but worsening after the treatment start date. TEAEs included both serious and non-serious TEAEs. Number of participants with TEAEs, Serious TEAEs and TEAEs leading to death were reported.
Time Frame: Up to 41 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cemiplimab 350 mg Q3W | Cemiplimab 350 mg Q3W + Ipilimumab 50 mg Q6W | Cemiplimab 1050 mg Q3W
Number analyzed (Participants) | 8 | 11 | 8
Participants
  Participants with any TEAE | 7 | 11 | 8
  Participants with any serious TEAE | 1 | 7 | 4
  Participants with any TEAE resulting in death | 0 | 2 | 1

6. Secondary Outcome: Number of Participants With Laboratory Test Abnormalities of Grade 2 or Higher Severity Based on National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) Grading System
Description: The laboratory measurements included hematology, chemistry, electrolytes and liver function. NCI-CTCAE was graded according to the following scale: Grade 1 (Mild): Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated; Grade 2 (Moderate): Moderate; minimal, local, or noninvasive intervention indicated; limiting age-appropriate instrumental Activities of Daily Living (ADL); Grade 3 (Severe): Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care ADL; Grade 4 (Life-threatening): Life-threatening consequences; urgent intervention indicated; Grade 5 (Death): Death related to AE.
Time Frame: Up to 41 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cemiplimab 350 mg Q3W | Cemiplimab 350 mg Q3W + Ipilimumab 50 mg Q6W | Cemiplimab 1050 mg Q3W
Number analyzed (Participants) | 8 | 11 | 8
Participants
  Hematology | 2 | 3 | 5
  Electrolytes | 3 | 3 | 1
  Liver Function | 2 | 3 | 1
  Chemistry | 1 | 1 | 0

ADVERSE EVENTS:
Time Frame: From first dose up to 41 months
Arm/Group | Cemiplimab 350 mg Q3W | Cemiplimab 350 mg Q3W + Ipilimumab 50 mg Q6W | Cemiplimab 1050 mg Q3W
All-Cause Mortality (participants affected / at risk) | 3/8 | 3/11 | 4/8
Serious Adverse Events (participants affected / at risk) | 1/8 | 7/11 | 4/8
Other Adverse Events (participants affected / at risk) | 7/8 | 11/11 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cemiplimab 350 mg Q3W (N=8) | Cemiplimab 350 mg Q3W + Ipilimumab 50 mg Q6W (N=11) | Cemiplimab 1050 mg Q3W (N=8)
Pneumonia (Infections and infestations) | 0 (0) | 3 (4) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Brain stem embolism (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Hemiparesis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Bradypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Cyanosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cemiplimab 350 mg Q3W (N=8) | Cemiplimab 350 mg Q3W + Ipilimumab 50 mg Q6W (N=11) | Cemiplimab 1050 mg Q3W (N=8)
Hypothyroidism (Endocrine disorders) | 0 (0) | 3 (3) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 2 (2) | 2 (2)
Hypophysitis (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 3 (3) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3) | 2 (5) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oral lichen planus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oral lichenoid reaction (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (3) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 3 (3) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 3 (3) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Fasciitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (4) | 2 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (5)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 2 (4) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0)
Dysarthria (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cauda equina syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 2 (2) | 0 (0)
Nervousness (Psychiatric disorders) | 0 (0) | 2 (3) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (2) | 3 (3) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Lichen planus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Skin odour abnormal (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Umbilical erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Eyelid ptosis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 3 (5) | 0 (0)
Asthenia (General disorders) | 2 (2) | 2 (5) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (2) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 2 (2)
Infusion site extravasation (General disorders) | 1 (1) | 0 (0) | 0 (0)
Oedema (General disorders) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (2) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood lactic acid increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood thyroid stimulating hormone decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 1 (1) | 1 (1)
Lipase increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Blood urea increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 4 (4) | 3 (6) | 3 (4)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 2 (2)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2)
Deafness (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Vestibular disorder (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Contrast media reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Pruritus genital (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Lymphoedema (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
All participants' tumors had PD-L1 expression levels of <50% at baseline. Therefore, the results do not present efficacy for participants with PD-L1 expression levels of ≥50% of tumor cells versus all participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator has the right to independently publish study results from the investigator's site after a multi-center publication, or a defined period after the completion of the study by all sites. The investigator must provide the sponsor a copy of any such publication derived from the study for review and comment in advance of any submission, and delay publication, if requested, to allow the Sponsor to preserve its proprietary rights.

DOCUMENTS (2):
  • Study Protocol (2018-05-01): https://cdn.clinicaltrials.gov/large-docs/63/NCT03430063/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-10): https://cdn.clinicaltrials.gov/large-docs/63/NCT03430063/SAP_001.pdf